CLINICAL TRIAL: NCT05920525
Title: Evaluation of Patient-reported Outcome Measures (PROMs) During Accelerating the En-masse Retraction of Upper Anterior Teeth Using a Low-intensity Direct Electrical Current: A Randomized Controlled Clinical Trial
Brief Title: Pain, Discomfort, and Acceptance During Using Electrical Stimulation to Accelerate Orthodontic Teeth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-11-2023
Record Dates: First submitted 2023-06-17; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Class II Malocclusion, Division 1
Keywords: Retraction of upper anterior teeth; Electrical stimulation; Coil springs
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical stimulation (Experimental): In this group of patients, retraction of upper anterior teeth will be done using backward traction, and the remodeling will be enhanced by very light electrical stimulation by a specific device.
  Interventions: Device: Electrical stimulation
- Traditional retraction of the front teeth (Active Comparator): In this group of patients, traditional traction of the front teeth will be employed without any acceleration method.
  Interventions: Procedure: Traditional retraction of the front upper teeth

INTERVENTIONS:
Device: Electrical stimulation — A specific device will be used to stimulate the remodeling procedures in the alveolar bone.
  Arms: Electrical stimulation
Procedure: Traditional retraction of the front upper teeth — The retraction will be performed using coil springs which will help in moving the anterior teeth backward without the need to employ any additional procedure or device to accelerate this movement.
  Arms: Traditional retraction of the front teeth

SUMMARY:
Forty patients with class II division 1 malocclusion who will require extraction of the upper first premolars as a part of the orthodontic treatment plan will be invited to participate in the study. They will be divided randomly into two groups: the electrical group and the control group. The en-masse retraction technique will be used to retract the upper anterior teeth using mini-implants as an anchor unit to provide the maximum anchorage and Nickle-Titanium closed coil springs that will be stretched from the mini-implants to the crimpable hooks on the base wire and applied 250 g of force per side.

A special removable electrical device will be used to provide electrical stimulation during the retraction phase.

The levels of pain and discomfort will be self-reported using a questionnaire with visual analog scales.

DETAILED DESCRIPTION:
Participants will be chosen from the patients attending the Department of Orthodontics in the Faculty of Dentistry at Damascus University. patients will be examined by the researcher, and any patient with class II division I malocclusion who meets the inclusion criteria will invite to participate in this trial. After giving them the information sheet, informed consent will be obtained from all patients who agreed to join the study.

Leveling and alignment will be performed using pre-adjusted fixed orthodontic appliances of 0.022 x 0.028-inch slot metal bracket with MBT prescription; the conventional wiring sequence will be followed until a 0.019 x 0.025 Stainless Steel base wire is attached.

The maxillary first premolars will be extracted, and skeletal anchoring will be applied before leveling and alignment will begin for all patients. self-drilling orthodontic mini-implants (diameter: 1.6 mm; length: 8 mm) will be placed between the roots of the maxillary second premolar and the first molar on each side.

The en-masse retraction will be done using Nickle-Titanium (NiTi) closed coil springs that stretched from crimpable hooks on the base wire to the mini-implants and applied 250 g of force per side. The force will be examined using a force gauge at every appointment (two weeks) until the completion of the retraction of the upper anterior (reaching a class I canine relationship and a correct incisor relationship).

A micro electrical current will be applied on the upper anterior teeth area using a removable intraorally device containing a small electrical circuit. Each patient in the experimental group will be asked to apply the electric accelerating device in the mouth for 5 hours daily.

The levels of pain and discomfort will be self-reported using a questionnaire with visual analog scales. 24 hours following the springs activation (T1), three days (T2), and one week (T3).

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy patients of both sexes
2. Age range: 17-25 years.
3. Class II Division 1 malocclusion:

   * Mild to moderate skeletal Class II (ANB = 5-7)
   * Protrusion less than 10 mm (5 to 10 mm of overjet)
   * Normal or vertical growth pattern (MM ≥ 26; SN-MP ≥ 33; Y Axis ≥ 65)
   * Dental crowding less than 3 mm
4. The presence of all permanent upper teeth (regardless of third molars).
5. Good oral and periodontal health:

   * Probing depth < 4 mm
   * No radiographic evidence of bone loss.
   * Gingival index ≤ 1
   * Plaque index ≤ 1

Exclusion Criteria:

1. Patients with previous orthodontic treatment.
2. Patients with severe skeletal dysplasia in all three dimensions.
3. Patients suffer from systemic diseases or syndromes
4. Patients on medication for systemic disorders, pregnancy, or steroid therapy.
5. Patients showing any signs of active periodontal disease

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Change in the perception of pain | Questionnaires will be filled at the following assessment times: at the 1st, 3rd, and 7th day of the first, second, and third months from the beginning of the en-masse retraction of upper anterior teeth
  Patients will be asked this question about their perception of pain. 'What is the degree of pain accompanying this moment?' Pain is assessed by asking the study participant to place a mark on a horizontal 100-mm line to indicate the level of pain being experienced. The left end of the line refers to no pain (VAS=0), whereas the right end refers to maximum (unimaginable) pain (VAS=100).
Change in the perception of discomfort | Questionnaires will be filled at the following assessment times: at the 1st, 3rd, and 7th day of the first, second, and third months from the beginning of the en-masse retraction of upper anterior teeth
  Patients will be asked this question about their perception of discomfort. 'What is the degree of discomfort that accompanies this moment?' Discomfort is assessed by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of discomfort being experienced. The left end of the line refers to no discomfort (VAS=0), whereas the right end refers to maximum (unimaginable) discomfort (VAS=100).

SECONDARY OUTCOMES:
Change in the perception of burning | Questionnaires will be filled at the following assessment times: at the 1st, 3rd, and 7th day of the first, second, and third months from the beginning of the en-masse retraction of upper anterior teeth
  Patients will be asked this question about their perception of burning. 'Do you feel any burning in the upper anterior teeth area?' burning is assessed by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of burning being experienced. The left end of the line refers to no burning (VAS=0), whereas the right end refers to maximum (unimaginable) burning (VAS=100).
Change in the perception of swelling | Questionnaires will be filled at the following assessment times: at the 1st, 3rd, and 7th day of the first, second, and third months from the beginning of the en-masse retraction of upper anterior teeth
  Patients will be asked this question about their perception of swelling. 'Do you feel any Swelling in the upper anterior teeth area?' Swelling is assessed by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of Swelling being experienced. The left end of the line refers to no Swelling (VAS=0), whereas the right end refers to maximum (unimaginable) Swelling (VAS=100).
Change in the chewing ability | Questionnaires will be filled at the following assessment times: at the 1st, 3rd, and 7th day of the first, second, and third months from the beginning of the en-masse retraction of upper anterior teeth
  Patients will be asked this question about their perception of chewing ability. 'what is the degree of chewing difficulties? ' difficulty in chewing is assessed by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of difficulty in swallowing being experienced. The left end of the line refers to no difficulty (VAS=0), whereas the right end refers to the maximum difficulty in mastication.
Change in the speech ability | Questionnaires will be filled at the following assessment times: at the 1st, 3rd, and 7th day of the first, second, and third months from the beginning of the en-masse retraction of upper anterior teeth
  Patients will be asked this question about their perception of speech ability. ''what is the degree of speech difficulties?' Difficulty in speech is assessed by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of difficulty in speech being experienced. The left end of the line refers to no difficulty (VAS=0), whereas the right end refers to maximum (unimaginable) difficulty (VAS=100).
Analgesic consumption | Questionnaires will be filled at the following assessment times: at the 1st, 3rd, and 7th day of the first, second, and third months from the beginning of the en-masse retraction of upper anterior teeth
  Patients will be asked this question about "Analgesic Consumption". 'Did you need to take pain analgesics?' Analgesic Consumption is assessed by asking the study participant about taking analgesics using a two-point scale (1. Yes, or 2. No).
Patients' satisfaction | Questionnaires will be filled at the end of the fifth month of the en-masse retraction
  Patients will be asked this question about satisfaction with orthodontic treatment.
  'How satisfied are you with your orthodontic treatment?' Satisfaction is assessed for both groups by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of satisfaction. The left end of the line refers to no satisfaction (VAS=0), whereas the right end refers to maximum satisfaction (VAS=100).
Ease of the procedure | Questionnaires will be filled at the end of the fifth month of the en-masse retraction
  Patients will be asked this question about the ease of the procedure. 'Was it getting used to the accelerating device? ' The procedure's easiness is assessed by asking the participant in the experimental group using a three-point scale (1. easy, 2. Medium, or 3. difficult).
The possibility of repeating the procedure | Questionnaires will be filled at the end of the fifth month of the en-masse retraction
  Patients will be asked this question about "The possibility of repeating the procedure.
  'Would you accept to undergo this treatment again?' Patients in the experimental group will be asked about the possibility of repeating the procedure if they can give their decision again. The answer will be collected using a two-point scale (1. Yes, or 2. No).
Recommendation of the procedure to a friend | Questionnaires will be filled at the end of the fifth month of the en-masse retraction
  Patients will be asked this question about the possibility of recommending the procedure to their friends.
  'Would you recommend a friend to undergo this treatment?' Patients in the experimental group will be asked if they would recommend this procedure to a friend. The answer will be collected using a two-point scale (1. Yes, or 2. No).

CONTACTS AND LOCATIONS:
Overall Officials: Rashad Ibrahim Shaadouh, DDS, Principal Investigator — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, University of Damsacus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roth PM, Thrash WJ. Effect of transcutaneous electrical nerve stimulation for controlling pain associated with orthodontic tooth movement. Am J Orthod Dentofacial Orthop. 1986 Aug;90(2):132-8. doi: 10.1016/0889-5406(86)90045-4. PMID 3488674
- [Background] Davidovitch Z, Finkelson MD, Steigman S, Shanfeld JL, Montgomery PC, Korostoff E. Electric currents, bone remodeling, and orthodontic tooth movement. II. Increase in rate of tooth movement and periodontal cyclic nucleotide levels by combined force and electric current. Am J Orthod. 1980 Jan;77(1):33-47. doi: 10.1016/0002-9416(80)90222-5. PMID 6243448
- [Background] Shaadouh RI, Hajeer MY, Al-Sabbagh R, Alam MK, Mahmoud G, Idris G. A Novel Method to Accelerate Orthodontic Tooth Movement Using Low-Intensity Direct Electrical Current in Patients Requiring en-Masse Retraction of the Upper Anterior Teeth: A Preliminary Clinical Report. Cureus. 2023 May 24;15(5):e39438. doi: 10.7759/cureus.39438. eCollection 2023 May. PMID 37234453
- [Derived] Shaadouh RI, Hajeer MY, Mahmoud GA, Almasri IA, Jaber ST, Alam MK. Patient-reported outcomes during accelerating the en-masse retraction of the upper anterior teeth using low-intensity electrical stimulation: a randomized controlled trial. Prog Orthod. 2024 May 13;25(1):17. doi: 10.1186/s40510-024-00517-3. PMID 38735912